CLINICAL TRIAL: NCT04771442
Title: Treatment With Stromal Vascular Fraction of Peyronie´s Disease in Humans
Brief Title: Stem Cell Treatment of Peyronie´s Disease.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-SVS
Record Dates: First submitted 2021-02-12; First posted 2021-02-25 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Penile Induration; Penile Diseases
Keywords: Stromal vascular fraction; Peyronie´s disease; Peyronie´s disease questionnaire; Erectile dysfunction
MeSH Terms: conditions — Penile Induration; Penile Diseases; Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stromal vascular fraction injection (Experimental): Intervention:
  Single injection with autologous adipose tissue-derived stromal vascular fraction cells in and around the plaque.
  Interventions: Drug: Stromal vascular fraction

INTERVENTIONS:
Drug: Stromal vascular fraction — Single dose
  Other Names: SVF

SUMMARY:
Purpose of the project is to investigate if a single injection of autologous stromal vascular fraction into and around plaque is a safe and suitable treatment.

Twentythree men > 18 years with Peyronie´s Disease in the chronic phase will be recruited.

The operative same-day procedure will be performed in general anaesthesia by a plastic surgeon. Before the patient wake, local anaesthesia is put around the penis. Processed stem cells are injected into the plaque/fibrosis subcutaneously.

There will be a follow up at 1, 3, 6, 12 months. It is a pilot study with no randomisation. The group will be compared to a historical control group.

ELIGIBILITY:
Inclusion Criteria:

1. Acquired penile curvature >30 and <90 degrees associated with a palpable penile plaque on physical examination.
2. One or several plaques at ultrasound screening.
3. Willingness to attend follow-up at 1, 3, 6 and 12 months.
4. Understand and speak Danish.
5. Men > 18 years of age

Exclusion Criteria:

Patients may not be:

1. Taking the medication Coumadin, Warfarin or NOAK (new oral anticoagulant).
2. Unable to achieve adequate erection with penile injection to access degree of curvature.
3. Undergoing definitive treatment for prostate cancer, bladder cancer, or other pelvic malignancies including surgery, external beam radiation therapy, brachytherapy, and cryotherapy.
4. With prior history of prostate cancer, hematologic disorders, chronic liver disease including cirrhosis and hepatitis C, disorders affecting the immune system, including infection with the human immunodeficiency virus, or psychiatric disorders including but not limited to major depression, schizophrenia, bipolar disease.
5. With a history of cerebrovascular incidents, a history of deep venous thrombosis within the past 5 years or a history of untreated or severe sleep apnoea.
6. With a clinically significant abnormal, results that would put the subject at increased risk or compromise the integrity of the study data, in the opinion of the investigator. Blood tests will be analysed for HIV, Hepatitis B and C and syphilis and those applicable within guidelines of the department.
7. Involved with any other projects with an investigational drug within 30 days.
8. In treatment for alcohol or drug abuse within six months.
9. With congenital deviation of penis.
10. Within six months treated with Collagenase, ESWT and/or other therapeutic injection in the plaque treatment for PD.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 22 (Actual)
Dates: Start 2022-09-09 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Change in the bend of the erect penis | [measured at baseline, 1, 3, 6, 12 months]
  Changes in degrees measured with a goniometer compared to baseline

SECONDARY OUTCOMES:
Change in Peyronie´s disease questionnaire bother symptoms | [measured at baseline, 1, 3, 6, 12 months]
  Will there be less bother symptoms compared to baseline? Score 0-44. The higher the score the more symptoms.
Change in International Index of Erectile Function score, | [measured at baseline, 1, 3, 6, 12 months].
  Score can be 5-25, the higher the score the less symptoms. Answers are compared to baseline.
Change in stretched Penile Length from symphysis to meatus of the glans (cm) | [measured at baseline, 1, and 12 months]
  Ruler
Change in penile Plaque size (mm3) | [measured at baseline, 1, and 12 months]
  Ultrasonic scanner

CONTACTS AND LOCATIONS:
Overall Officials: Majken Wiborg, MD, Principal Investigator — Hospital, Southwest Jytland
Locations (1):
- Sydvejstjysk Sygehus, Esbjerg, Denmark

IPD SHARING:
Plan to Share IPD: No